CLINICAL TRIAL: NCT00001437
Title: Trial of Pentoxifylline in Patients With Functional Disability Caused by Radiation-Induced Advanced Regional Fibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 950138; 95-C-0138
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 1999-05

CONDITIONS: Fibrosis; Radiation Injuries
Keywords: Cytokines; Fibrosis Intensity; Post-Radiation Fibrosis; Radiation Injury; Trental
MeSH Terms: conditions — Fibrosis; Radiation Injuries | interventions — Pentoxifylline

INTERVENTIONS:
Drug: pentoxifylline

SUMMARY:
After initial assessment of their condition by specified clinical and laboratory parameters, each of the patients will be treated for 8 weeks at the standard pentoxifylline dose (400 mg po TID). Objective and subjective response parameters will be re-assessed at the end of the treatment and 8 weeks later for possible decay of response.

DETAILED DESCRIPTION:
Patients with late fibrovascular sequelae of radiation or of combined radiation and surgery, with quantifiable symptomatology or disability, will be eligible for this trial. This protocol is designed as an open label one arm study. (A placebo controlled randomized trial was approved by the IRB but after extensive negotiation, drug and placebo in slow release formulation will not be provided by the manufacturer). Up to fifty patients will be recruited. After initial assessment of their condition by specified clinical and laboratory parameters, each of the patients will be treated for 8 weeks at the standard pentoxifylline dose (400 mg po TID). Objective and subjective response parameters will be re-assessed at the end of the treatment and 8 weeks later for possible decay of response.

In addition to symptomatic objective and subjective response, blood and urine will be collected for TNF, TGF-beta, and FGF. Cutaneous blood flow and collagen subtyping will be performed on a subset of patients using Laser Doppler, functional MRI techniques and subcutaneous tissue biopsies. We will examine for correlation between clinical response and these biological responses.

ELIGIBILITY:
POPULATION CHARACTERISTICS:

Regional advanced postradiation fibrosis of the neck, chest wall, pelvis, or extremities causing measurable impairment of specific function, i.e.: Decreased range of motion, Weakness, Sensory deficit, Pain requiring narcotics, Significantly altered activities of daily living.

None of these conditions present either before or during radiotherapy or attributed to surgery or chemotherapy.

Patients with prostate cancer allowed if prostate-specific antigen (PSA) is less than 4.0 ng/mL and the last 3 PSA values were stable or decreasing. Abnormal bone scan or film acceptable if consistent with degenerative disease.

No recurrent or metastatic cancer.

No concurrent second cancer.

PRIOR/CONCURRENT THERAPY: At least 3 months since pentoxifylline.

PATIENT CHARACTERISTICS:

Age: 18 and over.

Performance status: Karnofsky 70%-100% (unrelated to postradiation fibrosis).

CARDIOVASCULAR:

No symptomatic coronary artery disease with frequent anginal episodes necessitating any of the following during past 6 months: Coronary artery bypass, Angioplasty, Pacemaker placement, Thrombolytic treatment.

No chronic cardiac failure with persistent hemodynamic abnormality and ejection fraction less than 40%.

No coagulation, platelet, or vascular disorder that threatens to cause bleeding.

OTHER:

No intolerance to pentoxifylline or other xanthines (e.g., caffeine, theophylline, theobromine).

No seizure disorder.

No peptic ulcer disease.

Willing to undergo serial evaluations (excluding biopsies, laser Doppler, MRI) by NCI rehabilitation specialist for documentation and grading of functional disability.

No pregnant or nursing women.

Adequate contraception encouraged in fertile women.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50
Dates: Start 1995-06; Study Completion 2000-03

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States